CLINICAL TRIAL: NCT07064902
Title: Ivonescimab Combined With Chemoradiotherapy in High-Risk Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase II, Multicenter, Single-Arm Clinical Trial
Brief Title: Ivonescimab Combined With Chemoradiotherapy in High-Risk Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-113-FLK
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: PD-1/VEGF bispecific antibody; Chemoradiotherapy; Anti-PD-1 Therapy; Ivonescimab; Immunotherapy; Bispecific Antibody
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab arm (Experimental): Participants in this arm will receive induction chemotherapy with gemcitabine (1000 mg/m² on Days 1 and 8, Q3W × 3 cycles) and cisplatin (80 mg/m² on Day 1, Q3W × 3 cycles), combined with ivonescimab (10 mg/kg on Day 1, Q3W × 3 cycles). This will be followed by concurrent chemoradiotherapy (IMRT, 70 Gy/33 fractions, with cisplatin 100 mg/m² on Day 1, Q3W × 2 cycles), and then adjuvant ivonescimab monotherapy (10 mg/kg Q3W × 9 cycles).
  Interventions: Drug: Ivonescimab（AK112，a PD-1/VEGF bispecific antibody）

INTERVENTIONS:
Drug: Ivonescimab（AK112，a PD-1/VEGF bispecific antibody） — Ivonescimab (AK112) is a novel PD-1/VEGF bispecific antibody designed to simultaneously block PD-1-mediated immune evasion and inhibit VEGF-driven angiogenesis. In this study, ivonescimab is administered intravenously at a dose of 10 mg/kg every 3 weeks, starting on Day 1 of induction chemotherapy (3 cycles), followed by concurrent chemoradiotherapy (no ivonescimab), and then continued as adjuvant monotherapy for 9 additional cycles.

SUMMARY:
This trial aims to study the role of Ivonescimab combined with chemoradiotherapy in high-Risk locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The trial plans to enroll patients with T3N2M0+ Stage III (AJCC 9th) locoregionally advanced nasopharyngeal carcinoma (LANPC). Patients will receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin combined with ivonescimab, followed by concurrent chemoradiotherapy with cisplatin, and then 9 cycles of adjuvant ivonescimab. Ivonescimab will be administered every 3 weeks starting from day 1 of induction therapy and continued through the adjuvant phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years.
2. Histologically confirmed non-keratinizing carcinoma (according to WHO classification).
3. ECOG performance status of 0 or 1.
4. Previously untreated nasopharyngeal carcinoma staged as T3N2M0 or Stage III according to the AJCC 9th edition.
5. Adequate bone marrow function, defined as white blood cell count > 4×10⁹/L, hemoglobin > 90 g/L, and platelet count > 100×10⁹/L.
6. Adequate liver and renal function, defined as total bilirubin ≤ 1.5 × ULN; AST and/or ALT ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; and creatinine clearance ≥ 60 mL/min.
7. Normal thyroid function, amylase, lipase, pituitary function, inflammatory markers, myocardial enzymes, and ECG. For patients over 50 years old with a smoking history, pulmonary function test results must be normal. For patients with ECG abnormalities or a cardiovascular history not meeting exclusion criteria #8, echocardiography and cardiac function tests must be normal.
8. Signed informed consent and willingness to comply with all scheduled visits, treatment procedures, laboratory tests, and other study-related requirements.
9. Female participants of childbearing potential and male participants with female partners of childbearing potential must agree to use reliable contraception from screening until 1 year after completion of treatment.

Exclusion Criteria:

1. Tumor invasion of major blood vessels or significant recent (within 1 month) nasopharyngeal or nasal bleeding (>5 mL).
2. HBsAg positive with HBV DNA > 1×10³ copies/mL, or anti-HCV antibody positive.
3. HIV antibody positive or diagnosed with AIDS.
4. Active tuberculosis or history of active tuberculosis within the past year, unless adequately treated.
5. Active, known, or suspected autoimmune disease, including but not limited to uveitis, colitis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism, or asthma requiring bronchodilator therapy; exceptions include type 1 diabetes, hypothyroidism requiring hormone replacement, and localized skin conditions not requiring systemic therapy (e.g., vitiligo, psoriasis, or alopecia).
6. History of interstitial lung disease or pneumonitis requiring corticosteroid treatment within the past year.
7. Chronic systemic corticosteroid therapy (≥10 mg/day prednisone or equivalent) or use of other immunosuppressive therapy; inhaled or topical corticosteroids are allowed.
8. Uncontrolled cardiovascular disease, including NYHA Class ≥ 2 heart failure, unstable angina, myocardial infarction within 1 year, or supraventricular/ventricular arrhythmias requiring intervention.
9. Pregnant or breastfeeding women; pregnancy testing is required for women of childbearing potential.
10. History or presence of other malignancies, except adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, or papillary thyroid carcinoma.
11. Known hypersensitivity to monoclonal antibodies or any component of ivonescimab.
12. Active systemic infection requiring treatment within 1 week before study treatment.
13. Receipt of live vaccine within 30 days prior to the first dose of ivonescimab.
14. History of organ transplantation.
15. History of psychiatric illness, substance abuse, alcohol or drug dependence.
16. Any other condition which, in the opinion of the investigator, could compromise patient safety or compliance with the study protocol, including severe uncontrolled comorbidities, serious abnormal lab findings, or psychosocial risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | At the end of induction therapy
  Disappearance of all target lesions, with all pathological lymph nodes (including both target and non-target nodes) reduced in short axis to less than 10 mm.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the end of induction therapy
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve either a Complete Response (CR) or a Partial Response (PR) as assessed per RECIST v1.1 criteria.
Failure-free survival (FFS) | 2 years
  calculated from enrolment to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.
Overall survival (OS) | 2 years
  calculated from enrolment to the date of death from any cause.
Distant metastasis-free survival (DMFS) | 2 years
  calculated from enrolment to the date of first distant metastasis.
Locoregional recurrence-free survival (LRRFS) | 2 years
  calculated from enrolment to the date of locoregional persistence or 1st locoregional recurrence.
Adverse events (AEs) and serious adverse events (SAEs) | 2 years
  Analysis of adverse events (AEs) are based on treatmentrelated AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs.
  Graded according to CTCAE V5.0.
Quality of life (QoL) | 2 years
  Change in quality of life (QoL) will be assessed at six time points: prior to enrollment (baseline), after completion of induction immunotherapy, after completion of concurrent chemoradiotherapy, after the 5th cycle of adjuvant immunotherapy, after completion of all adjuvant immunotherapy, and at 6 months following the end of adjuvant immunotherapy. The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), version 3.0, will be used. This validated instrument contains 30 items, of which 24 are grouped into nine multi-item scales: five functional scales, three symptom scales, and one global health status/QoL scale. The remaining six items are single-item symptom scales. All 15 scales will be scored according to the EORTC QLQ-C30 Scoring Manual.Each scale is linearly transformed to a 0-100 scale. Higher scores indicate better functioning and QoL on functional and global health scales, but worse symptoms on symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated Hospital of Guilin Medical University, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto an online platform.

REFERENCES:
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Chen BJ, Chapuy B, Ouyang J, Sun HH, Roemer MG, Xu ML, Yu H, Fletcher CD, Freeman GJ, Shipp MA, Rodig SJ. PD-L1 expression is characteristic of a subset of aggressive B-cell lymphomas and virus-associated malignancies. Clin Cancer Res. 2013 Jul 1;19(13):3462-73. doi: 10.1158/1078-0432.CCR-13-0855. Epub 2013 May 14. PMID 23674495
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Wang J, Zhou C, Yao W, Wang Q, Min X, Chen G, Xu X, Li X, Xu F, Fang Y, Yang R, Yu G, Gong Y, Zhao J, Fan Y, Liu Q, Cao L, Yao Y, Liu Y, Li X, Wu J, He Z, Lu K, Jiang L, Hu C, Zhao W, Zhang B, Shi W, Zhang X, Cheng Y; CAPSTONE-1 Study Group. Adebrelimab or placebo plus carboplatin and etoposide as first-line treatment for extensive-stage small-cell lung cancer (CAPSTONE-1): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Jun;23(6):739-747. doi: 10.1016/S1470-2045(22)00224-8. Epub 2022 May 13. PMID 35576956
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573